CLINICAL TRIAL: NCT01783574
Title: Collaborative Study: Testosterone Antidepressant Augmentation in Women
Brief Title: Testosterone Antidepressant Augmentation in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Lawley Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012D000537; R34MH09931501A1 (Other: National Institute of Mental Health)
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Depression
Keywords: Depression; Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone (Active Comparator): Testosterone cream will be applied to skin for 8 weeks. Starting dose is 10 mg daily and will be titrated based on blood levels.
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): Placebo cream will appear identical to the testosterone cream and will be applied to skin for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone
  Other Names: AndroFeme 1(testosterone 1% w/v cream)
  Arms: Testosterone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators' hypotheses are: Low-dose testosterone augmentation improves depressive symptoms in women with Major Depressive Disorder (MDD) and antidepressant partial/nonresponse, adjunctive low-dose testosterone is safe and well-tolerated in women with MDD and antidepressant partial/nonresponse, and low-dose testosterone augmentation improves fatigue and sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age 21-75
2. Major depressive disorder including MADRS>/=12
3. Currently treated with an antidepressant monotherapy (1st, 2nd or 3rd trial in current episode), that has been taken at an adequate dose for at least six weeks.

Exclusion Criteria:

1. Serious suicide or homicide risk, as assessed by evaluating clinician
2. Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic
3. Substance use disorder active within last six months, or clinical suspicion of ongoing substance use disorder at the discretion of the study clinician at time of screening based on history and/or laboratory results.
4. Any history of psychotic features, bipolar disorder, or primary obsessive compulsive disorder, as assessed by SCID
5. Currently treated with typical or atypical antipsychotic medications, or lithium
6. Untreated hypothyroidism. If treated hypothyroidism, change in levothyroxine dose within the prior 3 mos
7. Use of androgens, including testosterone, dehydroepiandrosterone (DHEA) and methyltestosterone, within the prior three months
8. Any investigational psychotropic drug within the last thirty days
9. In the judgment of the study clinician, unlikely to be able to participate safely throughout the study period (three or more episodes of self-harm in the past year, documented history of poor treatment adherence, or frequent missed appointments (>50%) in the past year)
10. ALT > 3x upper limit of normal or creatinine> 3x upper limit
11. History of a hormone-responsive cancer

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Miller, MD, Principal Investigator — Massachusetts General Hospital; Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital; Linda L Carpenter, MD, Principal Investigator — Butler Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Dichtel LE, Carpenter LL, Nyer M, Mischoulon D, Kimball A, Deckersbach T, Dougherty DD, Schoenfeld DA, Fisher L, Cusin C, Dording C, Trinh NH, Pedrelli P, Yeung A, Farabaugh A, Papakostas GI, Chang T, Shapero BG, Chen J, Cassano P, Hahn EM, Rao EM, Brady RO Jr, Singh RJ, Tyrka AR, Price LH, Fava M, Miller KK. Low-Dose Testosterone Augmentation for Antidepressant-Resistant Major Depressive Disorder in Women: An 8-Week Randomized Placebo-Controlled Study. Am J Psychiatry. 2020 Oct 1;177(10):965-973. doi: 10.1176/appi.ajp.2020.19080844. Epub 2020 Jul 14. PMID 32660299

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone: Testosterone cream will be applied to skin for 8 weeks. Starting dose is 10 mg daily and will be titrated based on blood levels.
  Testosterone
- Placebo: Placebo cream will appear identical to the testosterone cream and will be applied to skin for 8 weeks.
  Placebo
Period: Overall Study
Arm/Group | Testosterone | Placebo
Started | 51 | 50
Completed | 46 | 41
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone | Placebo | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (14) | 48 (14) | 47 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 50 | 101
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 21 | 40
  Not Hispanic or Latino | 32 | 29 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 51 | 41 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.2 (7.6) | 30.3 (7.9) | 29.2 (7.8)
Mean MADRS Score [Mean (Standard Deviation); unit: units on a scale] — Montgomery-Asberg Depression Rating Score (MADRS) Score: This scale measures depression symptom severity. Higher scores indicate more severe depression symptom severity. The score range is 0-60 units on a scale.
  units on a scale | 26.8 (6.3) | 26.3 (5.4) | 26.6 (5.9)
Postmenopausal [Count of Participants; unit: Participants] | 20 | 26 | 46
Brief Fatigue Inventory [Mean (Standard Deviation); unit: units on a scale] — Brief Fatigue Inventory: This inventory measures fatigue severity. Higher scores indicate more severe fatigue. The range is 0-10 units on a scale.
  units on a scale | 6.2 (1.9) | 5.6 (2.0) | 5.9 (2.0)
Derogatis Inventory of Sexual Function [Mean (Standard Deviation); unit: units on a scale] — Derogatis Interview of Sexual Function (Total Score): This scale measures sexual function. Lower scores indicate worse sexual function. The score range for this questionnaire is 0-160.
  units on a scale | 32.8 (27.3) | 38.7 (30.1) | 35.7 (28.7)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptom Severity
Description: Montgomery-Asberg Depression Rating Score (MADRS) Score: This scale measures depression symptom severity. Higher scores indicate more severe depression symptom severity. The score range is 0-60 units on a scale.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 51 | 50
units on a scale | 15.3 (1.4) | 14.1 (1.4)

2. Secondary Outcome: Fatigue
Description: Brief Fatigue Inventory: This inventory measures fatigue severity. Higher scores indicate more severe fatigue. The range is 0-10 units on a scale.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 51 | 50
units on a scale | 4.0 (0.3) | 3.7 (0.4)

3. Secondary Outcome: Sexual Dysfunction
Description: Derogatis Interview of Sexual Function (Total Score): This scale measures sexual function. Lower scores indicate worse sexual function. The score range for this questionnaire is 0-160.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 51 | 50
units on a scale | 45.1 (4.7) | 47.5 (5.4)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Definition of serious adverse event is as defined on the clinicaltrials.gov website.
Arm/Group | Testosterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 15/51 | 13/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone (N=51) | Placebo (N=50)
Acne (Skin and subcutaneous tissue disorders) | 7 | 3
Hot flashes (Reproductive system and breast disorders) | 2 | 6
Headache (General disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT01783574/Prot_002.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT01783574/SAP_003.pdf